CLINICAL TRIAL: NCT01761383
Title: Nintendo Wii and Schizophrenia. A Pilot Study.
Brief Title: Role of Nintendo Wii in Improving Negative Symptoms and Quality of Life in Chronic Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Walmart (Industry)
Responsible Party: Principal Investigator, Dr. Martin Feakins, Prinicpal Investigator, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6006092
Record Dates: First submitted 2012-11-01; First posted 2013-01-04 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Schizophrenia
Keywords: Chronic Schizophrenia; Nintendo Wii; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nintendo Wii and Chronic Schizophrenia (Experimental): Participants enrolled in the study will be provided with the Nintendo Wii console and Nintendo Wii Fit Plus video games to use for the duration of the study (6 months) with no restrictions or limitations on the games participants are allowed to play or duration of play. There will be 5 home visits over a 6-month period to evaluate Nintendo Wii use and assess patients'health, functioning and quality of life with the use of self report questionnaires and psychiatric assessment.
  Interventions: Other: Nintendo Wii video console and Nintendo Wii Fit Plus games

INTERVENTIONS:
Other: Nintendo Wii video console and Nintendo Wii Fit Plus games — The intervention will be provision of Nintendo Wii console and Wii Fit Plus video games to use for the duration of the study with no restrictions or limitations on the games participants are allowed to play or duration of play. There will be 5 home visits over a 6-month period to evaluate Nintendo Wii use and assess patients'health, functioning and quality of life.

SUMMARY:
The purpose of this study is to determine whether the use of Nintendo Wii will help improve negative symptoms of Schizophrenia and quality of life of patients with chronic Schizophrenia.

DETAILED DESCRIPTION:
The proposed study seeks to determine whether any benefit in daily functioning and quality of life can be gained from using the Nintendo Wii video game console in chronic mental illness, namely schizophrenia. There is a small research base on the use of the Wii console in elderly nursing home residents as a means of increasing mobility, with attendant benefits in areas such as falls, quality of life, and relief of subsyndromal depression. For individuals with schizophrenia, adjunct exercise therapy has been associated with gains in both psychiatric and physical symptoms. However, people with schizophrenia face physical and functional barriers in initiating and continuing organized activity programs. Thus, the Nintendo Wii Fit Plus interactive fitness video game is being proposed as a novel way of introducing and engaging people with schizophrenia in various forms of physical activity.

As the first study to assess the use of the Nintendo Wii in chronic mental illness, the purpose of this pilot study is to assess the feasibility and the capacity of the Nintendo Wii in improving the health and functioning of people with severe, chronic schizophrenia. Although it is hypothesized that Nintendo Wii use will lead to gains in these domains, the information gained from this study will be used to determine specific areas of benefit and to assess whether any observed differences in outcome measures are sufficient to warrant a full-scale study. Furthermore, this initial study aims to pilot the interview schedule, clarify wording on the questionnaires, ensure that all important areas have been covered by the questionnaires, and determine whether participants are capable of meeting the demands of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Schizophrenia defined by the DSM-IV-TR (Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition-Text Revision)
* Males or females aged 18 years of older
* Participate in the Community High Intensity Treatment Team (CHITT) out-patient program
* Certified by their physician to participate in physical activity

Exclusion Criteria:

* History of violence or other risks that may endanger study research assistants during home visits

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Quality of life. | 6 months
  To assess whether any benefit in daily functioning and quality of life can be gained from using the Nintendo Wii video game console in people with chronic Schizophrenia. Assessed with the use of Short Form (36 questions)self report Health Survey (SF-36), Global Assessment of Functioning (GAF) Scale and the Clinical Global Impression-Schizophrenia(CGI-SCH)Scale.

SECONDARY OUTCOMES:
Weight. | 6 months
  To assess whether the use of Nintendo Wii will help in weight reduction [assessed using Body Mass Index (BMI) calculations and weight measurements] in patients with Chronic Schizophrenia.
Subjective overall functioning. | 6 months
  To assess whether the use of Nintendo Wii will help to: reduce cigarette consumption, improve subjective quality of life and motivation [assessed using a self report Visual Analog Scale(VAS)] in patients with Chronic Schizophrenia.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Feakins, M.D., Principal Investigator — Department of Psychiatry at Queen's University, Kingston, Ontario, Canada
Locations (1):
- Community High Intensity Treatment Team (CHITT) at Providence Care Mental Health Services, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No